CLINICAL TRIAL: NCT03216590
Title: Can Preoperative Compressive Draping Reduce Soft Tissue Swelling During Shoulder Arthroscopy? A Prospective Randomized Trial
Brief Title: The Effect of Draping on Swelling in Shoulder Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HYMC-17-0033
Record Dates: First submitted 2017-07-09; First posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Shoulder Arthroscopy; Soft Tissue Swelling
Keywords: Shoulder Arthroscopy; Soft Tissue Swelling; Rotator Cuff Repair; Shoulder Arthroscopy Complications

STUDY DESIGN:
Intervention Model Description: After signing an informed consent participants will be randomised to one of the two study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard draping (No Intervention): Shoulder arthroscopy will be performed using standard draping with the shoulder exposed.
- Compressive draping (Experimental): After standard preparation similar to the no-intervention group, the shoulder will be draped with compressive draping using adhesive incise drape (Ioban™2 Antimicrobial Incise Drape, 3M Inc.,USA)
  Interventions: Device: Compressive draping using adhesive incise drape

INTERVENTIONS:
Device: Compressive draping using adhesive incise drape — In the intervention group the shoulder will be drape with compressive draping using adhesive incise drape (Ioban™2 Antimicrobial Incise Drape, 3M Inc.,USA).
  Arms: Compressive draping

SUMMARY:
Strategies to minimize soft tissue swelling during shoulder arthroscopy are constantly sought after. The investigators propose an unfamiliar method which may reduce tissue swelling during shoulder arthroscopy.

DETAILED DESCRIPTION:
Fluid extravasation into the surrounding tissue is common in shoulder arthroscopy. It frequently leads to soft tissue swelling and edema which results in poor visualization and prolonged surgical time. While usually resolves uneventfully within 12 hours, excessive fluid extravasation into the soft tissue around the shoulder may lead to serious consequences and complications such as airway compromise, tracheal deviation, neuropraxias, habdomyoloysis and skin necrosis have been reported in the literature. Methods aimed at reducing soft tissue swelling during shoulder arthroscopy in order to avoid complications (e.g., low pump pressure, short arthroscopic time) are routinely practiced. Nevertheless, fluid extravasation and soft tissue swelling remains a concern in shoulder arthroscopy.

The purpose of the current study is to evaluate whether applying local compression to the shoulder by preoperative compressive draping will reduce soft tissue swelling during shoulder arthroscopy. To the investigators' knowledge, no previous study evaluated the influence of applying compressive draping to the shoulder on soft tissue swelling in shoulder arthroscopy.

ELIGIBILITY:
Inclusion criteria for the study are defined as:

1. Surgery indicated for chronic symptomatic RC tear unresponsive to non-operative treatment over a minimal period of 6 months.
2. Small to medium size tears (<3 cm).
3. Age older than 18 years.
4. ASA score 1or 2.
5. Body mass index (BMI) < 35.
6. Willingness to provide an informed consent.

Exclusion criteria:

1. Pregnant women.
2. Arthroscopic procedure that was converted to an open ("mini-open") surgery.
3. Patients who do not meet the above mentioned inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-07-20 (Estimated); Primary Completion 2017-12-20 (Estimated); Study Completion 2017-12-20 (Estimated)

PRIMARY OUTCOMES:
Change on shoulder circumference | Immediate post-operative
  The change in shoulder circumference will be assessed at the end of the procedure. Shoulder circumference before and at the end of the procedure will be measured from the mid-point between the coracoid process and anterior axillary fold anteriorly to the mid-point between the scapular spine and the posterior axillary fold posteriorly.

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Uri, Principal Investigator — Hillel Yaffe Medical Center

REFERENCES:
- [Derived] Uri O, Alfandari L, Yaron R, Kettanie A, Laufer G, Behrbalk E. Effect of Compressive Shoulder Draping With Adhesive Incise Drape on Soft Tissue Swelling in Shoulder Arthroscopy: A Prospective Randomized Trial. Orthop J Sports Med. 2024 Feb 19;12(2):23259671241229736. doi: 10.1177/23259671241229736. eCollection 2024 Feb. PMID 38379580